CLINICAL TRIAL: NCT02518334
Title: Wine Consumption and Glycemic Control
Acronym: WGC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Wine and GC
Record Dates: First submitted 2012-02-08; First posted 2015-08-07 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type two diabetes; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alcohol consumption (Experimental): Alcohol consumption and wine consumption
  Interventions: Other: Alcohol consumption

INTERVENTIONS:
Other: Alcohol consumption — 28 grams (2 drinks) of ethanol will be consumed either in the form of wine or vodka.

SUMMARY:
Many studies have reported that alcoholic beverage consumption, especially in the form of wine, reduces the risk of developing type 2 diabetes by as much as 40%. This association suggests that wine consumption may somehow improve the body's ability to control its blood glucose concentration. Indeed, it has been reported that when wine is consumed immediately prior to ingestion of glucose, the release of insulin is enhanced and blood glucose concentration is lowered. The mechanism of wine's effects on blood glucose concentration is unknown, but is likely related to its ethanol or antioxidant content. In this study, the investigators plan to test whether wine or plain ethanol (vodka) ingestion alters the control of blood glucose in subjects who have diabetes or pre-diabetes.

DETAILED DESCRIPTION:
Our central hypothesis is that improvement in glycemic control by acute consumption of wine is mediated by ethanol. Subjects will have type 2 diabetes, pre-diabetes, and be sedentary and obese (BMI >30). Subjects' glycemic control will be assessed by an oral glucose tolerance test (OGTT) at three different time points. One OGTT will occur shortly after consumption of red wine, the second after consumption of vodka containing the identical amount of ethanol as the wine treatment, and the third OGTT will occur shortly after consumption of an equal volume of water. The three OGTTs will be administered in random order.

ELIGIBILITY:
Inclusion Criteria:

* insulin resistant: diagnosed with pre-diabetes or fasting blood glucose >/= 97 mg/dL
* T2D: diagnosed by primary care physician
* at risk of type 2 diabetes (obesity and physically inactive)
* age: 21-65

Exclusion Criteria:

* smoking
* insulin use (other than once daily)
* physically active (>30 mins aerobic exercise two days/week)
* recent (>3 mo) changes in medication use or dose
* uncontrolled type two diabetes (HbA1C >10%)
* advanced retinopathy or neuropathy
* pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Oral glucose tolerance test | 3 weeks
  Measurement of blood glucose taken every 15 minutes over a course of three hours.

CONTACTS AND LOCATIONS:
Overall Officials: John P Thyfault, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avogaro A, Watanabe RM, Dall'Arche A, De Kreutzenberg SV, Tiengo A, Pacini G. Acute alcohol consumption improves insulin action without affecting insulin secretion in type 2 diabetic subjects. Diabetes Care. 2004 Jun;27(6):1369-74. doi: 10.2337/diacare.27.6.1369. PMID 15161790